CLINICAL TRIAL: NCT01141101
Title: Risk Factors for Early Infant Colonization With Methicillin-Resistant Staphylococcus Aureus
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Stephen Pelton, BMC Faculty, Boston Medical Center
Other Study IDs: H-29160
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Methicillin-resistant Staphylococcus Aureus
Keywords: Methicillin-resistant Staphylococcus aureus; Neonatal; Vertical transmission; Horizontal transmission; MRSA colonization in enrolled infants; MRSA colonization obtained from maternal source; MRSA colonization obtained from source other that mother

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — MRSA isolates from the nose, axilla or perineum from mothers, infants and house hold contacts and caregivers enrolled in the study will be retained only for the duration of the study for use in molecular analysis for the purpose of this study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MRSA-exposed: The MRSA-exposed group will include 100 MRSA-colonized mothers and their babies
- MRSA-unexposed: The MRSA-unexposed group will include 100 MRSA-negative mothers and their babies.

SUMMARY:
The prevalence of Methicillin-resistant Staphylococcus aureus (MRSA) colonization and infections have been increasing in the general population, including the pediatric population. It has been reported that MRSA colonization persists for up to four years, and therefore the youngest pediatric patients, specifically those who are less than 2 years of age, have a high risk of prolonged colonization during a period of time when they are susceptible to significant skin and soft tissue infections (SSTIs) attributable to MRSA. Once prolonged colonization takes place, recurrent SSTIs are commonplace, resulting in substantial morbidity and in some cases mortality, as well as a significant cost to the healthcare system. Individuals colonized with MRSA have an increased risk of developing MRSA infections, which range from mild disease, such as carbuncles, to severe infections, such as necrotizing pneumonia and toxic shock syndrome. The prevalence of severe MRSA infections is also greatest in neonates and infants, where increased MRSA colonization has been observed. In the early infant period, the most common manifestation of MRSA disease is pustular skin lesions, which affect approximately 5% of the general population, with MRSA-colonization being a major risk factor for this disease. Moreover, the prevalence of pustular disease is increasing in the general population, and there are numerous case reports of invasive, life-threatening MRSA disease in the early infant period.

Corresponding to the increasing prevalence in the community, the carriage of MRSA in pregnant women has also escalated, and vaginal carriage is significant in pregnant women. As an analogy, maternal vaginal Group B Streptococcal (GBS) colonization is the major risk for infant colonization regardless of whether early or late neonatal colonization or disease occurs. It is quite feasible that vaginal MRSA carriage predisposes newborns to colonization during the birthing process; however, this mechanism has not yet been well studied. There are other mechanisms implicated for early infant colonization, including close contact with MRSA-colonized mothers through daily care and breastfeeding. MRSA colonization in one household member greatly predisposes colonization in others; therefore, early infant colonization could result from contact with other MRSA-colonized individuals in a household. Currently, it is not clear which factors are the most important in influencing early infant MRSA colonization and subsequent infection.

Not only is the prevalence of MRSA colonization and infection on the rise, but there have been few if any measures that have been established to prevent colonization and subsequent infection in adults and children. Eradication measures have shown limited long-term benefit. If vertical transmission of MRSA can be established as a critical event in the pathogenesis of disease, potentially effective strategies could be tested, and possibly the spread of MRSA in the community interrupted.

Hypotheses and Specific Aims:

1. Identify the proportion, rate and time of MRSA colonization in infants born to mothers with and without MRSA colonization;
2. Compare risk factors for infant MRSA colonization in these two groups;
3. Determine the prevalence and risk factors for developing MRSA infections in the MRSA-colonized infant.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at > 32 weeks of gestation.
* Mother must have been tested for MRSA prior to birth.
* Mother must be willing to provide informed consent for herself and infant.
* Mothers feel household contacts and caregivers will be willing to enroll in the study.
* Household contacts must be willing to provide informed consent (if greater than 18 years of age) or parent of household contact must be willing to provide informed consent for minors and the minor must provide assent (if greater than age 7) to enroll in study.
* Infant care givers must be willing to provide informed consent (if greater than 18 years of age) or parent of infant care giver must be willing to provide informed consent for minors and the minor must provide assent (if greater than age 7) to enroll in study.

Exclusion criteria:

* Infants born at < 32 weeks gestation.
* Infants who will not be receiving their primary care at Boston Medical Center.
* Household contact or Infant Care giver not willing to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The exposed group will include 100 MRSA-colonized mothers and their babies. The unexposed group will include 100 MRSA-negative mothers and their babies. The groups will be conveniently selected from all mothers and infants meeting the inclusion and exclusion criteria each month. Enrollment will continue until 100 babies and mothers in the MRSA-positive mother group and 100 babies and mothers in MRSA-negative mother group are enrolled. We estimate that enrollment will require approximately 18 months to complete.
  Household contacts of infants will be enrolled. A contact is defined as any individual who had or has had the same primary residences (who has lived in the same house for at least one week) as the infant since the infant's birth. We will ask the infants mother to identify the infants household contacts.
  Infant care givers include any person who provides daily care to infant for at least 4 hours per day at least 3 days of week.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
We will compare infants' MRSA-positivity rates in the exposed versus the unexposed study groups. | 18 months

SECONDARY OUTCOMES:
We will determine if infant MRSA positivity appears earlier in exposed infants versus unexposed infants. | 18 months
For infants who become MRSA-positive we will determine if their strain of MRSA is the same as their mothers' or other household contacts or care giver who is determined to be MRSA-positive. | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States